CLINICAL TRIAL: NCT07216092
Title: The Role of Audio-recorded Gut-hypnotherapy on Sleep Disturbance, Sleep-related Impairment and Abdominal Pain in Pediatric Functional Abdominal Pain Disorders
Brief Title: Audio-recorded Gut-Hypnotherapy for Sleep and Pain in Pediatric Abdominal Pain Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital at Montefiore (Other)
Responsible Party: Principal Investigator, Lily Barash, Physician, Children's Hospital at Montefiore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14317
Record Dates: First submitted 2025-09-17; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Irritable Bowel Syndrome; Disorders of Gut-brain Interaction
Keywords: gut-directed hypnotherapy; disorders of gut-brain interaction; irritable bowel syndrome; sleep-related impairment; sleep disturbance
MeSH Terms: conditions — Irritable Bowel Syndrome; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gut-directed hypnotherapy (Experimental): 6-week series of audio-recorded sessions of gut-directed hypnotherapy
  Interventions: Other: Gut-directed Hypnotherapy
- Standard Medical Therapy (No Intervention): This group continued their usual medical care for 6 weeks

INTERVENTIONS:
Other: Gut-directed Hypnotherapy — Gut-directed hypnotherapy is an evidence-based treatment that combines hypnosis with therapeutic suggestions that target the gut-brain connection. Through relaxation, imagery, and suggestions, patients learn to better control their pain.
  Arms: Gut-directed hypnotherapy

SUMMARY:
Children with irritable bowel syndrome (IBS) and functional abdominal pain- not otherwise specified (FAP-NOS) have higher rates of poor sleep quality. This can be associated with worse abdominal pain and quality of life, but few treatments target sleep. Gut-directed hypnotherapy (GDH) has been shown to reduce abdominal pain and has been hypothesized to improve sleep, but this has not been studied. This study investigates the use of a home-based audio program of GDH as a feasibility intervention for children and whether it can also help with sleep quality. Children aged 8-18 with IBS or FAP-NOS were enrolled from three children's hospitals. Participants in one group completed 6 weeks of GDH sessions at home. Sleep, abdominal pain, and daily functioning were tracked through online surveys. Participants in the control group continued their usual medical care first, and then crossed over into the GDH program.

DETAILED DESCRIPTION:
Children with pain-predominant disorders of gut-brain interaction (DGBI) including irritable bowel syndrome (IBS) and functional abdominal pain-not otherwise specified (FAP-NOS) frequently experience sleep-related impairment, which is linked to increased pain severity, functional disability, and health care utilization. Gut-directed hypnotherapy (GDH) is an evidence-based treatment for pediatric DGBI that has been hypothesized to improve sleep, although this has not been studied. This pilot randomized controlled trial evaluates the feasibility of implementing a 6-week, audio-guided GDH program at home and explores effect sizes for sleep, abdominal pain, quality of life, and anxiety outcomes. Children ages 8-18 meeting Rome IV criteria for IBS or FAP-NOS and at least mild sleep disturbance or sleep impairment were recruited virtually from three pediatric gastroenterology centers. Participants were randomized to either standard medical therapy (SMT) or GDH; SMT participants crossed over to GDH after 6 weeks. Primary outcomes were feasibility as measured by adherence, interest, and satisfaction and sleep effect size. Secondary exploratory aims included abdominal pain, functional disability, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* ages 8 to 18 years
* met Rome IV criteria for FAP-NOS or IBS
* abdominal pain severity >3/10 in the past 2 weeks
* minimum of 1 day of pain in the past 2 weeks
* mild SRI and/or SD as determined by the PROMIS 4- question short-form questionnaires
* stable medication regimen or dietary therapy for >2 weeks prior to enrollment

Exclusion Criteria:

* disability that could hinder their understanding of the audio material
* previous experience with guided imagery for treatment of abdominal pain
* psychiatric disorder with psychotic elements such as dissociative symptoms
* other chronic gastrointestinal disease including inflammatory bowel disease, celiac disease, or eosinophilic esophagitis
* other chronic inflammatory conditions
* previous gastrointestinal surgery
* a diagnosis of a sleep disorder such as narcolepsy or sleep apnea.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of adherence and satisfaction to hypnotherapy treatment protocol | This was assessed throughout the 6 week course by completion of daily abdominal pain surveys and at the end of the 6 week hypnotherapy course.
  Feasibility was measured through treatment adherence and participant satisfaction. Adherence was measured by number of pre-audio surveys completed and self-reported number of audios completed per week. A 5-point likert scale was used to determine enrolled participant satisfaction with hypnotherapy at the end of the intervention.
Treatment effect size for Sleep Quality as measured by PROMIS Questionnaire for sleep-related impairment and sleep disturbance | enrollment to the end of the 3-month follow up period
  Patient- reported outcomes measurement information system (PROMIS) sleep related impairment and sleep disturbance surveys were used to measure sleep quality. This scale produces T-scores ranging from about 25-75, normalized to a population mean of 50 and a standard devision of 10. For this measure, a higher T-score indicates a greater severity of sleep related impairment or sleep disturbance.

SECONDARY OUTCOMES:
Abdominal pain | enrollment to the end of the 3-month follow up period
  Defined as pain severity and frequency. Assessed using numerical modified abdominal pain index. Frequency and intensity scores were multiplied to yield a combined score with possible range of 0 to 50. Daily abdominal pain was assessed using Faces pain Scale- reviewed, rating pain from 0-10.
Functional disability | enrollment to the end of the 3-month follow up period
  Disability is assessed and defined by the Functional Disability Inventory tool. This is a numerical tool, resulting in a total score that ranges from 0 to 60. A higher total score indicates greater degree of functional disability.
Anxiety | enrollment to the end of the 3-month follow up period
  Patient- reported outcomes measurement information system (PROMIS) emotional distress-- anxiety was used to measure anxiety. This scale produces T-scores ranging from about 25-75, normalized to a population mean of 50 and a standard devision of 10. For this measure, a higher T-score indicates a greater severity of anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Borlack, Principal Investigator — Montefiore
Locations (1):
- Children's Hospital at Montefiore, Mahwah, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
It is a small sample size, this will risk privacy and confidentiality for participants

REFERENCES:
- [Background] van Tilburg MA, Chitkara DK, Palsson OS, Turner M, Blois-Martin N, Ulshen M, Whitehead WE. Audio-recorded guided imagery treatment reduces functional abdominal pain in children: a pilot study. Pediatrics. 2009 Nov;124(5):e890-7. doi: 10.1542/peds.2009-0028. Epub 2009 Oct 12. PMID 19822590
- [Background] Groen J, Gordon M, Chogle A, Benninga M, Borlack R, Borrelli O, Darbari A, Dolinsek J, Khlevner J, Di Lorenzo C, Person H, Sanghavi R, Snyder J, Thapar N, Vlieger A, Sinopoulou V, Tabbers M, Saps M. ESPGHAN/NASPGHAN guidelines for treatment of irritable bowel syndrome and functional abdominal pain-not otherwise specified in children aged 4-18 years. J Pediatr Gastroenterol Nutr. 2025 Aug;81(2):442-471. doi: 10.1002/jpn3.70070. Epub 2025 May 30. PMID 40444524
- [Background] Palsson OS, van Tilburg M. Hypnosis and Guided Imagery Treatment for Gastrointestinal Disorders: Experience With Scripted Protocols Developed at the University of North Carolina. Am J Clin Hypn. 2015 Jul;58(1):5-21. doi: 10.1080/00029157.2015.1012705. PMID 26046714
- [Background] Mamoune S, Mener E, Chapron A, Poimboeuf J. Hypnotherapy and insomnia: A narrative review of the literature. Complement Ther Med. 2022 May;65:102805. doi: 10.1016/j.ctim.2022.102805. Epub 2022 Jan 21. PMID 35074550
- [Background] Rutten JMTM, Vlieger AM, Frankenhuis C, George EK, Groeneweg M, Norbruis OF, Tjon A Ten W, van Wering HM, Dijkgraaf MGW, Merkus MP, Benninga MA. Home-Based Hypnotherapy Self-exercises vs Individual Hypnotherapy With a Therapist for Treatment of Pediatric Irritable Bowel Syndrome, Functional Abdominal Pain, or Functional Abdominal Pain Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2017 May 1;171(5):470-477. doi: 10.1001/jamapediatrics.2017.0091. PMID 28346581
- [Background] Vasant DH, Hasan SS, Cruickshanks P, Whorwell PJ. Gut-focused hypnotherapy for children and adolescents with irritable bowel syndrome. Frontline Gastroenterol. 2020 Nov 23;12(7):570-577. doi: 10.1136/flgastro-2020-101679. eCollection 2021. PMID 34917314
- [Background] Gulewitsch MD, Muller J, Hautzinger M, Schlarb AA. Brief hypnotherapeutic-behavioral intervention for functional abdominal pain and irritable bowel syndrome in childhood: a randomized controlled trial. Eur J Pediatr. 2013 Aug;172(8):1043-51. doi: 10.1007/s00431-013-1990-y. Epub 2013 Apr 9. PMID 23568514
- [Background] Santucci NR, Velasco-Benitez CA, Velasco-Suarez DA, King C, Byars K, Dye T, Li J, Saps M. Youth With Functional Abdominal Pain Disorders Have More Sleep Disturbances. A School-Based Study. Neurogastroenterol Motil. 2025 Apr;37(4):e14992. doi: 10.1111/nmo.14992. Epub 2024 Dec 31. PMID 39737536
- [Background] Haim A, Pillar G, Pecht A, Lerner A, Tov N, Jaffe M, Hardoff D. Sleep patterns in children and adolescents with functional recurrent abdominal pain: objective versus subjective assessment. Acta Paediatr. 2004 May;93(5):677-80. PMID 15174794
- [Background] Huntley ED, Campo JV, Dahl RE, Lewin DS. Sleep characteristics of youth with functional abdominal pain and a healthy comparison group. J Pediatr Psychol. 2007 Sep;32(8):938-49. doi: 10.1093/jpepsy/jsm032. Epub 2007 Jul 12. PMID 17627965
- [Background] Patel A, Hasak S, Cassell B, Ciorba MA, Vivio EE, Kumar M, Gyawali CP, Sayuk GS. Effects of disturbed sleep on gastrointestinal and somatic pain symptoms in irritable bowel syndrome. Aliment Pharmacol Ther. 2016 Aug;44(3):246-58. doi: 10.1111/apt.13677. Epub 2016 May 30. PMID 27240555
- [Background] Murphy LK, Palermo TM, Tham SW, Stone AL, Han GT, Bruehl S, Garber J, Walker LS. Comorbid Sleep Disturbance in Adolescents with Functional Abdominal Pain. Behav Sleep Med. 2021 Jul-Aug;19(4):471-480. doi: 10.1080/15402002.2020.1781634. Epub 2020 Jun 23. PMID 32573267
- [Background] Schurman JV, Friesen CA, Dai H, Danda CE, Hyman PE, Cocjin JT. Sleep problems and functional disability in children with functional gastrointestinal disorders: an examination of the potential mediating effects of physical and emotional symptoms. BMC Gastroenterol. 2012 Oct 15;12:142. doi: 10.1186/1471-230X-12-142. PMID 23067390
- [Background] Thapar N, Benninga MA, Crowell MD, Di Lorenzo C, Mack I, Nurko S, Saps M, Shulman RJ, Szajewska H, van Tilburg MAL, Enck P. Paediatric functional abdominal pain disorders. Nat Rev Dis Primers. 2020 Nov 5;6(1):89. doi: 10.1038/s41572-020-00222-5. PMID 33154368

DOCUMENTS (1):
  • Informed Consent Form (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT07216092/ICF_000.pdf